CLINICAL TRIAL: NCT05256901
Title: Effectiveness of Sugammadex Versus Neostigmine on Neuromuscular Reversal in Pediatric Patients Undergoing Laparoscopic Appendectomy for Acute Appendicitis: A Randomized Controlled Trial
Brief Title: Sugammadex vs Neostigmine Reversal in Pediatric Appendectomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was terminated due to lack of funding.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Laura Gilbertson, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00003913
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Results first posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Appendicitis; Surgery
Keywords: laparoscopic
MeSH Terms: conditions — Appendicitis | interventions — Sugammadex; Neostigmine; Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sugammadex (Experimental): The reversal agent, Sugammadex, will be administered at the start of closure.
  Interventions: Drug: Sugammadex
- Neostigmine/Glycopyrrolate (Active Comparator): The reversal agent, Neostigmine, will be administered at the start of closure.
  Interventions: Drug: Neostigmine/Glycopyrrolate

INTERVENTIONS:
Drug: Sugammadex — Participants will receive 4mg/kg for a TOF 0-1 and 2mg/kg for a train of four (TOF) 2 or more.
  Other Names: Intervention Group
  Arms: Sugammadex
Drug: Neostigmine/Glycopyrrolate — Participants will receive 0.07mg/kg of Neostigmine and 0.01mg/kg of Glycopyrrolate, administered by anesthesia once at least two twitches are present.
  Other Names: Regular Care
  Arms: Neostigmine/Glycopyrrolate

SUMMARY:
This study is designed as a randomized controlled trial with patients assigned to neuromuscular reversal with either sugammadex or neostigmine/glycopyrrolate reversal. The study will not be blinded to the anesthesiologist to allow for appropriate decision-making on timing and dosage of reversal. This is a single-center study.

DETAILED DESCRIPTION:
Patients presenting to the operating room for laparoscopic appendectomy with a diagnosis of acute appendicitis require rapid sequence induction (RSI) due to significant vomiting and concern for increased gastric content. For this reason, succinylcholine-accompanied by neostigmine-is predominantly used in adults for RSI to prevent potential aspiration. Unfortunately, in pediatric patients, there are many concerns about the use of succinylcholine, including complications such as bradycardia, hyperkalemia, dysrhythmias, and cardiac arrest from undiagnosed skeletal muscle myopathy. For many anesthesiologists, these concerns prompted the decision to use a non-depolarizing muscle relaxant such as rocuronium for induction. However, if the standard RSI dose is used, it often results in residual paralysis at the end of short procedures such as laparoscopic appendectomies. It has recently been demonstrated that prolonged paralysis is prevalent even at low doses of rocuronium in pediatric patients. For these reasons, it is imperative to find a way to provide adequate and safe

RSI conditions for intubation, appropriate muscle relaxation for laparoscopic procedures, and the ability to quickly reverse neuromuscular blockade in this pediatric population. Sugammadex has the potential to allow for the utilization of an appropriate RSI dose of rocuronium for intubation, as it provides the ability to reverse neuromuscular blockade earlier than the neostigmine reversal, which is currently the standard of care. Retrospective reviews have shown the use of Sugammadex in pediatric patients to be safe and effective. However, there has not been prospective data about the effect on operating room efficiency of brief pediatric procedures such as laparoscopic appendectomies, one of the most common urgent pediatric surgeries performed. There are numerous other potential benefits of using sugammadex over typical reversal, including the quicker return of bowel function, faster time to tolerance of an oral diet, and decreased exposure to volatile anesthesia. The return of bowel function is particularly important in pediatric patients undergoing laparoscopic procedures. The research team hypothesizes that the utilization of sugammadex in pediatrics results in a quicker return to bowel function. This has previously been demonstrated in adults, but data are lacking in the pediatric population. Researchers also hypothesize that patients receiving sugammadex versus neostigmine reversal will have an improved time to tolerance of an oral diet, which may impact wound healing and nutrition. As anesthesiologists often underdose rocuronium in these short procedures, due to a lack of quick reversal options, high levels of volatile anesthesia are utilized to compensate for inadequate muscle relaxation. With the use of sugammadex allowing for proper muscle relaxation throughout the entire case, researchers hypothesize that patients will have a lower total volatile anesthetic exposure during the procedure. This is exceedingly important in pediatric anesthesia, where the detrimental effects of volatile anesthetics on the developing brain have been demonstrated in numerous animal studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients 2-17 years of age
* Diagnosis of acute appendicitis
* Patient undergoing laparoscopic appendectomy at Children's Healthcare of Atlanta- Egleston.
* Parent or Legal Authorized Representative willing to participate, able to understand and sign an informed consent

Exclusion Criteria:

* Patient with an allergy to Sugammadex or Neostigmine
* History of renal dysfunction
* Parent or legal guardian unwilling or unable or unable to understand the informed consent

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Gilbertson, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team will share Individual participant data that underlie the results (text, tables, figures, and appendices) reported in the article, after the deidentification
Supporting Information: Study Protocol, SAP
Time Frame: The research team will share the data immediately following publication and ending 3 years following article publication.
Access Criteria: Proposals should be directed to laura.gilbertson@emory.edu. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Groups:
- Sugammadex: The reversal agent, Sugammadex, will be administered at the start of closure.
  Sugammadex: Participants will receive 4mg/kg for a TOF 0-1 and 2mg/kg for a train of four (TOF) 2 or greater.
Period: Overall Study
Arm/Group | Sugammadex | Neostigmine/Glycopyrrolate
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex | Neostigmine/Glycopyrrolate | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 11 | 22
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.55 (3.50) | 10.18 (3.52) | 11.37 (3.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 7 | 5 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 5 | 5 | 10
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Total Time From Surgery End to Out of the Operating Room (OR)
Description: The time from the end of surgery to discharge from the OR will be evaluated via the Epic computer chart after discharge from the hospital.
Time Frame: Up to 2 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex | Neostigmine/Glycopyrrolate
Number analyzed (Participants) | 11 | 11
minutes | 9.55 (3.03) | 10.82 (4.87)

2. Secondary Outcome: Total Time to First Bowel Movement
Description: Time to first bowel movement will be evaluated via the Epic computer record after discharge from the hospital
Time Frame: Up to 48 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Sugammadex | Neostigmine/Glycopyrrolate
Number analyzed (Participants) | 11 | 11
hours | 18.4 (6.7) | 23.78 (16.74)

3. Secondary Outcome: Total Time to Tolerance of an Oral Diet
Description: The research team will evaluate via the Epic computer record after discharge from the hospital
Time Frame: Up to 24 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Sugammadex | Neostigmine/Glycopyrrolate
Number analyzed (Participants) | 11 | 11
hours | 4.3 (1.96) | 8.05 (6.75)

4. Secondary Outcome: Total Time of Inhalational Anesthesia Exposure
Description: evaluated via the Epic computer record after discharge from the hospital
Time Frame: Up to 5 hours (depending on length of surgical procedure)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex | Neostigmine/Glycopyrrolate
Number analyzed (Participants) | 11 | 11
minutes | 121.30 (40.14) | 142.94 (34.32)

5. Secondary Outcome: Length of Stay in the Post-anesthesia Care Unit (PACU)
Description: PACU length of stay was evaluated via the Epic computer record after discharge from the hospital
Time Frame: Up to 5 hours (on average depending on post anesthesia recovery)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex | Neostigmine/Glycopyrrolate
Number analyzed (Participants) | 11 | 11
minutes | 27.91 (9.07) | 37.73 (12.65)

6. Secondary Outcome: Hospital Length of Stay (LoS)
Description: Hospital LoS will be evaluated via the Epic computer record after discharge from the hospital
Time Frame: Up to 5 days (depending on length of hospitalization)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Sugammadex | Neostigmine/Glycopyrrolate
Number analyzed (Participants) | 11 | 11
hours | 34.64 (39.07) | 49.51 (50.56)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected from the time of consent to participate in the study up to hospital discharge, with an average duration of up to five (5) days.
Arm/Group | Sugammadex | Neostigmine/Glycopyrrolate
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-25): https://cdn.clinicaltrials.gov/large-docs/01/NCT05256901/Prot_SAP_000.pdf